CLINICAL TRIAL: NCT02528292
Title: Phase 4 Study of Clinical Disease Activity and Modulation of Synovial Lymphoid Structures and B Cell Function in Patients With Rheumatoid Arthritis Undergoing Treatment With Anti-TNF Therapy
Brief Title: Clinical Disease Activity and Modulation of Synovial Lymphoid Structures and B Cell Function in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UCB-007275
Record Dates: First submitted 2011-08-05; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-TNF; Ultrasound; Synovial histomorphology; Ectopic Lymphoneogenesis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial tissue and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Rheumatoid Arthritis: Patients with active Rheumatoid Arthritis with a DAS 28 score of greater than 5.1 and eligible for anti-TNF alpha therapy according to National Institute for Clinical Excellence guidelines will be recruited in this study
  Interventions: Procedure: Synovial biopsy; Drug: Anti-TNF therapy

INTERVENTIONS:
Procedure: Synovial biopsy — Ultrasound guided synovial biopsy of inflamed joint
Drug: Anti-TNF therapy — Therapy will include, but not limited to Etanercept, Certolizumab Pegol, Adalimumab and Infliximab

SUMMARY:
This study will be an open label observational prospective study assessing the clinical efficacy of antiTNFα therapy and the alteration/impact on the synovial tissue, with specific regard to lymphoid aggregation, over a period of 12 months in patients with rheumatoid arthritis.

Rheumatoid arthritis (RA) is one of the most important chronic inflammatory disorders in the UK. It affects approximately 1% of adults and causes considerable morbidity, substantially reduces quality of life and has a significant mortality. It results in large direct medical costs as well as extensive indirect social costs. Despite the significant therapeutic progress following the introduction of antiTNFα, a cure for RA is still elusive. At present the reasons for the variation in clinical response are not known. The main aim of this study is to test the hypothesis that there are distinct molecular and cellular phenotypes present within the synovial tissue that define specific disease subsets and provide characteristic prognostic implications. In particular, the aim is to assess the relationship between the presence of ectopic lymphoneogenesis (ELN) within the rheumatoid synovial membrane and response to antiTNFα therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 and ≤ 75 years of age, with RA as defined by the 1987 revised ACR classification criteria.
* Patients must fulfill the National Institute for Clinical Excellence guidelines for TNF Blocking Therapy in RA.
* Patients must be on MTX for at least 4 months, with a stable dose of 7.525 mg/week for a minimum of 4 weeks.
* Men and women of childbearing potential must use adequate birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study.
* Patients must be able to adhere to the study visit schedule.
* Patients must be capable of giving informed consent and the consent must be obtained prior to any screening procedures.
* Must have a chest Xray within 3 months prior to commencement of antiTNFα with no evidence of malignancy, infection or fibrosis.

Exclusion Criteria:

* Women who are pregnant or breast feeding.
* Use of any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Previous use of antiTNF biologics.
* Treatment with any other therapeutic agent targeted at reducing TNF (eg, pentoxifylline, thalidomide, etc.) within 3 months of screening.
* Serious infections (such as, HIV, HBV, pneumonia or pyelonephritis) in the previous 3 months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
* Have active TB or have evidence of latent TB (old or latent TB on chest Xray, without adequate therapy for TB initiated prior to first dose of study drug). Also excluded are patients with evidence of an old or latent TB infection without documented adequate therapy.
* Presence of a transplanted organ (with the exception of a corneal transplant >3 months prior to screening).
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Known recent substance abuse (drug or alcohol).
* Poor tolerability of venepuncture required blood sampling during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within Rheumatology secondary care services with active Rheumatoid Arthritis will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of change in synovial ectopic lymphoneogenesis with EULAR response criteria using DAS28 | Baseline and 12 months

SECONDARY OUTCOMES:
Disability and health status assessed using the HAQ questionnaire | Baseline and 12 months
X-ray progression | Baseline and 12 months
  Progression of x-ray damage of hand and feet using modified van der heidje / sharp score
Change in synovial histomorphology with treatment | baseline and 3 months
Correlation of peripheral blood lymphocytes including, Treg markers and, B cell subsets | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Costantino Pitzalis, MD, PhD, Principal Investigator — Barts and the London NHS Trust
Locations (1):
- Rheumatology Department, Mile End Hospital, Barts and The Royal London NHS Trust, London, London, United Kingdom